CLINICAL TRIAL: NCT04655118
Title: A Phase 2 Multicenter Study of TL-895 in Subjects With Relapsed/Refractory Myelofibrosis, Janus Kinase Inhibitor Intolerant Myelofibrosis, Janus Kinase Inhibitor Treatment Ineligible Myelofibrosis, or Indolent Systemic Mastocytosis
Brief Title: Study of TL-895 in Subjects With Myelofibrosis or Indolent Systemic Mastocytosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TL-895-201
Record Dates: First submitted 2020-11-24; First posted 2020-12-07 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Myelofibrosis; Indolent Systemic Mastocytosis
MeSH Terms: conditions — Primary Myelofibrosis; Mastocytosis, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Cohort 1a, Relapsed/Refractory Myelofibrosis (Experimental): 150 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 1b, Relapsed/Refractory Myelofibrosis (Experimental): 300 mg of TL-895 will be administered orally, once daily (QD) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 1c, Relapsed/Refractory Myelofibrosis (Experimental): 300 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 1d, Relapsed/Refractory Myelofibrosis (Experimental): 450 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 2a, JAKi Intolerant Myelofibrosis (Experimental): 150 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 2b, JAKi Intolerant Myelofibrosis (Experimental): 300 mg of TL-895 will be administered orally, once daily (QD) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 3a, JAKi Ineligible Myelofibrosis with platelet count of ≥ 25 and < 50 × 109/L (Experimental): 150 mg of TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 3b, JAKi Ineligible Myelofibrosis with platelet count of ≥ 25 and < 50 × 109/L (Experimental): 300 mg of TL-895 will be administered orally, once daily (QD) continuously starting on Day 1 in a 28-day cycle.
  Interventions: Drug: TL-895
- Cohort 5a, Indolent Systemic Mastocytosis (Experimental): TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle in combination with best supportive care (BSC).
  Interventions: Drug: TL-895
- Cohort 5b, Indolent Systemic Mastocytosis (Experimental): TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle in combination with BSC.
  Interventions: Drug: TL-895
- Cohort 5c, Indolent Systemic Mastocytosis (Experimental): TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle in combination with BSC.
  Interventions: Drug: TL-895
- Cohort 5d, Indolent Systemic Mastocytosis (Experimental): TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle in combination with BSC.
  Interventions: Drug: TL-895
- Cohort 5e, Indolent Systemic Mastocytosis (Placebo Comparator): Placebo to match TL-895 will be administered orally, twice daily (BID) continuously starting on Day 1 in a 28-day cycle in combination with BSC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TL-895 — TL-895 is an experimental tyrosine kinase inhibitor drug taken by mouth.
  Arms: Cohort 1a, Relapsed/Refractory Myelofibrosis; Cohort 1b, Relapsed/Refractory Myelofibrosis; Cohort 1c, Relapsed/Refractory Myelofibrosis; Cohort 1d, Relapsed/Refractory Myelofibrosis; Cohort 2a, JAKi Intolerant Myelofibrosis; Cohort 2b, JAKi Intolerant Myelofibrosis; Cohort 3a, JAKi Ineligible Myelofibrosis with platelet count of ≥ 25 and < 50 × 109/L; Cohort 3b, JAKi Ineligible Myelofibrosis with platelet count of ≥ 25 and < 50 × 109/L; Cohort 5a, Indolent Systemic Mastocytosis; Cohort 5b, Indolent Systemic Mastocytosis; Cohort 5c, Indolent Systemic Mastocytosis; Cohort 5d, Indolent Systemic Mastocytosis
Drug: Placebo — Placebo to match TL-895
  Arms: Cohort 5e, Indolent Systemic Mastocytosis

SUMMARY:
This study evaluates TL-895, a potent, orally-available and highly selective irreversible tyrosine kinase inhibitor for the treatment of Myelofibrosis (Cohorts 1-3) or Indolent Systemic Mastocytosis (Cohort 5). Participants must be diagnosed with Myelofibrosis and be relapsed/refractory (e.g., having failed prior therapy), intolerant, or ineligible to receive JAKi treatment, or be diagnosed with Indolent Systemic Mastocytosis.

ELIGIBILITY:
Cohorts 1-3

Key Inclusion Criteria:

* Adults ≥18 years of age
* Confirmed diagnosis of PMF, post-PV MF, or post-ET MF, as assessed by treating physician according to the World Health Organization (WHO) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
* Adequate hematologic, hepatic, and renal functions
* MF symptoms as defined by having at least 2 symptoms with an average baseline (Day -7 to Day -1) score of at least 1 for each of the 2 symptoms per MFSAF v4.0
* Cohort 3 only: Ineligibility for JAKi treatment with a platelet count of ≥ 25 and < 50 x 10^9/L

Key Exclusion Criteria:

* Prior treatment with any BTK or BMX inhibitors
* Prior treatment with JAKi within 28 days prior to study treatment
* Prior splenectomy or splenic irradiation within 24 weeks prior to first dose of study treatment

Cohort 5

Key Inclusion Criteria:

* Adults ≥18 years of age
* Confirmed diagnosis of ISM as defined by WHO diagnostic criteria based on review of bone marrow biopsy pathology report results
* Subject must have moderate-to-severe symptoms

Key Exclusion Criteria:

* Prior treatment with any BTK or BMX inhibitors
* Prior treatment with Avapritinib, bezuclastinib, or BLU-263/elenestinib
* Diagnosis with another myeloproliferative disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1-3: Determine the RP2D of TL-895 | 9 months
  The RP2D for Cohorts 1, 2 and 3 will be reported
Cohort 5: Determine the RP2D of TL-895 | Week 24
  The RP2D for Cohort 5 will be reported

SECONDARY OUTCOMES:
Cohorts 1-3: Spleen volume reduction (SVR) rate | Week 24
  The proportion of subjects achieving ≥35% SVR at Week 24 by MRI or CT scan (central review).
Cohort 5: Changes in patient reported symptoms | Week 12
  Mean change in patient reported symptom assessment

CONTACTS AND LOCATIONS:
Locations (52):
- United States (6):
  - University of Colorado - Aurora Cancer Center, Aurora, Colorado
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Gabrail Cancer Center, Canton, Ohio
  - University of Cincinnati (UC) Physicians Company, LLC, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Border Medical Oncology, East Albury
  - Southern Oncology Specialists, Kogarah
  - Royal Perth Hospital, Perth
  - St Vincent's Hospital Sydney, Sydney
- Belgium (2):
  - Chu De Liège, Liège
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Instituto de Estudos e Pesquisas Sao Lucas - IEP - Sao Lucas, São Paulo, Brazil
- Bulgaria (2):
  - University Hospital "St Ivan Rilski", Sofia
  - Military Medical Academy, Sofia
- France (3):
  - CH Le Mans, Le Mans
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - CHU de Nice - Hopital L' Archet II, Nice
- Germany (5):
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Marien Hospital Duesseldorf, Düsseldorf
  - Klinik fur Innere Medizin IV - Hamatologie/Onkologie, Universitatsklinikum Hall, Halle
  - Universitaetsklinikum Jena, Jena
  - Praxisklinik fur Hamatologie und Onkologie, Koblenz
- Hungary (4):
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Szabolcs-Szatmár-Bereg Megyei Önkormányzat Jósa András Oktatókórház Megyei-Városi Tüdőgondozó Intézete, Nyíregyháza
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Italy (9):
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico-San Marco - Presidio Ospedaliero G. Rodolico, Catania
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Maggiore Della Carita', Novara
  - Azienda Ospedaliera di Perugia-Ospedale S. Maria della Misericordia, Perugia
  - AUSL della Romagna-Ospedale S.Maria delle Croci, Ravenna
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Reggio Calabria
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
- Poland (4):
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Klinika Hematologi, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk
  - Klinika Hematologii Collegium Medicum Uniwersytetu Jagiellonskiego, Krakow
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Klinika Hematologii, Nowotworów Krwi i Transplantacji Szpiku, Wroclaw
- South Korea (3):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
- Spain (5):
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Salamanca University Hospital, Salamanca
  - Hospital Quirónsalud Zaragoza, Zaragoza
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei